CLINICAL TRIAL: NCT07268456
Title: Volumetric Bone Reconstruction of Complex Alveolar Ridge Defects Using CAD/CAM-Customized Titanium Meshes: A Retrospective Study
Brief Title: Treatment of Complex Ridge Defects With Custom Meshes
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Duygu Kilic, Principal Investigator, TC Erciyes University
Other Study IDs: EU2025/64
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Bone Defects
Keywords: Alveolar ridge augmentation; CAD/CAM; Customized titanium mesh; Guided bone regeneration; Mesh exposure; Volumetric analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- custom mesh group: All operations were performed under local anesthesia (4% articaine with 1:100,000 epinephrine). A mid-crestal incision with vertical releasing incisions was made, and full-thickness buccal and lingual/palatal flaps were elevated. Decortication was applied to enhance vascularization. Bone harvesting was performed from the mandibular ramus using bone scrapers.
  Autogenous bone was mixed 1:1 with deproteinized bovine bone (Tutobone, Tutogen Medical GmbH). The graft was inserted into the custom mesh, which was then secured over the defect using titanium screws. Grafting was completed through mesh openings until full volume was achieved. The mesh was covered with a resorbable collagen membrane, and primary closure was obtained with tension-free sutures

SUMMARY:
Brief introduction: After tooth extraction, alveolar defects may hinder implant placement. Digital imaging and CAD/CAM advances allow creation of patient-specific titanium meshes for effective bone augmentation.

Objective: This study aimed to evaluate the clinical effectiveness of customized titanium meshes produced using computer-aided design and manufacturing (CAD/CAM) technologies in the horizontal and vertical augmentation of complex alveolar ridge defects prior to implant placement.

DETAILED DESCRIPTION:
Implant dentistry is a recognized and dependable method for restoring functionality and aesthetics in individuals with partial or total tooth loss. Following tooth loss or extraction, the alveolar bone undergoes gradual resorption and atrophy. This process generally commences with a notable horizontal decrease in ridge width over the initial six months, succeeded by vertical bone loss over time. Consequently, patients often have horizontal, vertical, or mixed alveolar defects that hinder later implant implantation.

Attaining sufficient bone volume before implant surgery is essential for enduring functional and aesthetic results. Horizontal and vertical bone augmentation procedures have demonstrated efficacy in enhancing alveolar ridge dimensions and facilitating the outcome of implant therapy. Among them, guided bone regeneration (GBR) is one of the most extensively utilized and evidence-based techniques, due to its reliability and capacity to facilitate new bone creation. Guided Bone Regeneration (GBR) employs resorbable or non-resorbable membranes alongside bone graft materials to safeguard the clot, prevent soft tissue encroachment, and promote osteogenesis within the defect.

Notwithstanding its prevalent application, the choice of membrane type continues to be a subject of contention. Resorbable membranes are manageable; nonetheless, they may exhibit inadequate mechanical stability, which could jeopardize the volume of regenerated bone. Conversely, non-resorbable membranes, especially titanium-reinforced polytetrafluoroethylene (PTFE) membranes, demonstrate enhanced space maintenance and they are considered more reliable for addressing extensive flaws.

In the late 1960s, titanium meshes were offered as a substitute for conventional membranes. These meshes provide improved stiffness and biocompatibility, rendering them appropriate for intricate ridge augmentation scenarios. Nevertheless, conventional titanium meshes require manual adjustment during surgery, potentially prolonging operative time and resulting in problems such as soft tissue dehiscence, mesh exposure, and postoperative infection due to inadequate fit.

Recent advancements in digital imaging and CAD/CAM technology have facilitated the creation of patient-specific titanium meshes, tailored according to preoperative cone beam computed tomography (CBCT) data. These bespoke meshes provide enhanced anatomical conformity, decrease intraoperative handling, reduce surgery duration, and mitigate problems linked to conventional meshes. Their smooth surface and exact fit to the bone defects correlate with reduced exposure rates and improved surgical results. However, limited studies have quantitatively assessed the volumetric outcomes of CAD/CAM-fabricated meshes using standardized CBCT-based protocols.

This study aims to assess the clinical and radiological effects of employing customized titanium meshes for alveolar ridge augmentation in individuals with horizontal and/or vertical bone defects. Key outcomes encompass bone volume increase, exposure rates, and the overall viability of the surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Comprised the presence of alveolar bone defects involving both vertical and horizontal components in edentulous regions of the maxilla.
* Comprised the presence of alveolar bone defects involving both vertical and horizontal components in edentulous regions of the mandible.

Exclusion Criteria:

* uncontrolled systemic disease,
* poor oral hygiene,
* active oral infections,
* autoimmune or inflammatory oral diseases,
* pregnancy,
* histories of head and neck radiotherapy, chemotherapy in the past six months,
* corticosteroid use,
* or smoking more than 10 cigarettes per day.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective study included all patients who underwent bone augmentation using customized titanium meshes at the Department of Periodontology, Faculty of Dentistry, Erciyes University, between July 2022 and June 2024.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
planned bone volume | beginning to 4-6 months
  planned bone volume when mesh was designed
planned horizontal width | beginning to 4-6 months
  planned horizontal width when mesh was designed
planned vertical height | beginning to 4-6 months
  planned vertical height when mesh was designed
regenerated bone volume | beginning to 4-6 months
  regenerated bone volume when mesh was applied to the patient
regenerated horizontal width | beginning to 4-6 months
  regenerated horizontal width when mesh was applied to the patient
regenerated vertical height | beginning to 4-6 months
  regenerated vertical height when mesh was applied to the patient

SECONDARY OUTCOMES:
mesh exposure rate | begining to 4-6 months
  the number of exposed titanum mesh

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Kilic, Asst. prof., Principal Investigator — Erciyes Uni
Locations (1):
- Erciyes University, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy and ethical restrictions.